CLINICAL TRIAL: NCT00865891
Title: A Relative Bioavailability Study of 60 mg Nifedipine Extended Release Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R05-0099
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Nifedipine; Healthy subjects
MeSH Terms: interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Nifedipine Extended Release tablets 60 mg, single dose
  Interventions: Drug: Nifedipine Extended Release tablets 60 mg, single dose
- B (Active Comparator): ADALAT® CC Extended Release Tablets 60 mg
  Interventions: Drug: ADALAT® CC Extended Release Tablets 60 mg

INTERVENTIONS:
Drug: Nifedipine Extended Release tablets 60 mg, single dose — A: Experimental Subjects received Abrica Pharmaceuticals LLLP formulated products under fasting conditions
  Other Names: Nifedipine
  Arms: A
Drug: ADALAT® CC Extended Release Tablets 60 mg — B: Active comparator Subjects received Bayer Pharmaceuticals Corporation, Bayer HealthCare formulated products under fasting conditions
  Other Names: Nifedipine
  Arms: B

SUMMARY:
The purpose of this study is to compare the relative bioavailability of Nifedipine ER tablets 60 mg by Abrica Pharmaceuticals LLLP with that of ADALAT® CC Extended Release Tablets 60 mg by Bayer Pharmaceuticals Corporation, Bayer HealthCare following a single oral dose (1 x 60 mg tablet) in healthy adult volunteers under fasting conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, single dose, two-way crossover study under fasting conditions

Official Title: A Relative Bioavailability Study of 60 mg Nifedipine Extended Release tablets Under Fasting Conditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers selected for this study will be healthy men and women 18 to 45 years of age inclusive at the time of dosing. The weight range will not exceed ± 20% for height and body frame as per Desirable Weights for Adults -1983 Metropolitan Height and Weight Table.
* Screening Procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems.
* The screening clinical laboratory procedures will include:

  * HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential; RBC count, platelet count;
  * CLINICAL CHEMISTRY: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase;
  * HIV antibody and hepatitis B surface antigen screens;

    •*URINALYSIS: by dipstick, microscopic examination if dipstick positive; and.
  * URINE DRUG SCREEN: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates and phencyclidine.
  * SERUM PREGNANCY SCREEN (female volunteers only)
* If female and:

  * of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s) condom with spermicide, diaphragm with sperriIicide, intrauterine device. (IUD), or abstinence; or
  * is postmenopausal for at least I year; or
  * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the medical investigator).
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Volunteers demonstrating a positive hepatitis B surface antigen, hepatitis C antibody or HIV antibody.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are currently breastfeeding.
* Volunteers with a history of allergic response(s) to nifedipine or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the medical investigator).
* Volunteers who currently use tobacco products.
* Volunteers who have taken any drug known to induce or inhibit hepatic• drug metabolism in the 28 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
* Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Volunteers who report receiving any investigational drug within 28 days prior to Period I dosing.
* Volunteers who report taking any systemic prescription medication in the 14 days prior to Period I dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2005-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 60 hours

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson,, Pharm.D,, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States